CLINICAL TRIAL: NCT05946460
Title: Neoadjuvant Aumolertinib in Patients With AI-diagnosed EGFR-mutant High-risk Pulmonary Ground-glass Opacity: A Single-arm, Phase II Trial
Brief Title: Neoadjuvant Aumolertinib in Patients With AI-diagnosed EGFR-mutant High-risk Pulmonary Ground-glass Opacity.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CATO-2301
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer
Keywords: Aumolertinib; Neoadjuvant Treatment; AI-diagnosed; EGFR-mutant; Ground-glass Opacity
MeSH Terms: conditions — Lung Neoplasms | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Aumolertinib (Experimental): Single Arm
  Interventions: Drug: Aumolertinib

INTERVENTIONS:
Drug: Aumolertinib — Aumolertinib treatment (110mg, p.o., QD) for 8 weeks

SUMMARY:
This is a prospective, single-center, single-arm, phase II study evaluating the efficacy and safety of neoadjuvant aumolertinib in previously untreated patients with AI-diagnosed EGFR-mutant and resectable pulmonary ground-glass opacity.

After informed consent signed, enrolled patients will undergo a treatment period and a follow-up period. During the treatment period, patients will receive aumolertinib treatment (110mg, p.o., QD) for 8 weeks. The surgery can be performed after a 1 to 2-week discontinuation period; if the patient does not consent to undergo surgery, follow-up can be conducted instead. If patients experience disease progression during the treatment period, they will be withdrawn from the study. During the follow-up period, the investigator will provide appropriate treatment recommendations based on the patient's condition and pathological results after surgical resection of the target lesion. Postoperative patients (or patients who completed the medication treatment and were followed up) will be monitored every six months for a duration of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 years old (including 18) and 75 years old (including 75).
2. No prior history of receiving anti-tumor treatment.
3. Presence of at least one resectable malignant EGFR-mutant pulmonary ground-glass nodule diagnosed by AI (CTR ≤ 0.5, EGFR mutation prediction value ≥ 0.82), with a nodule diameter between 0.8-3cm (including both 0.8cm and 3cm).
4. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1.
5. Adequate function of important organs, as follows:

   1. Bone marrow: Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L, platelets ≥ 100 × 10^9/L, hemoglobin ≥ 9 g/dl.
   2. Liver: Bilirubin ≤ 1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 times ULN.
   3. Kidney: Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 ml/min.
6. Female of childbearing potential must use appropriate contraceptive measures during the study and should not be breastfeeding for at least 3 months after discontinuation of study treatment. Before initiation of treatment, a negative pregnancy test is required, or one of the following criteria should be met to demonstrate no risk of pregnancy:

   1. Postmenopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
   2. Women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the institution.
   3. Previously undergone irreversible surgical sterilization, including hysterectomy, bilateral oophorectomy, or bilateral salpingectomy (except for bilateral tubal ligation).
7. Male patients should use barrier contraception (i.e., condoms) from enrollment until 3 months after discontinuation of study treatment.
8. Voluntary participation of the subject and signed informed consent.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Diagnosis or treatment of any other malignant tumor within the past 5 years (excluding patients with previously resected basal cell carcinoma of the skin or other in situ cancers).
2. Use of systemic anti-tumor treatment, including chemotherapy, radiotherapy, or targeted therapy (including but not limited to monoclonal antibodies, small molecule tyrosine kinase inhibitors), before the study enrollment.
3. Prediction of benign nodules or EGFR wild-type after AI tool assessment of the target lesion.
4. Patient's organ system conditions:

   1. History of interstitial lung disease, drug-induced interstitial disease, radiation pneumonitis requiring steroid treatment, or any clinically active interstitial lung disease.
   2. Evidence of interstitial lung disease detected on baseline CT scan.
   3. Evidence of severe or uncontrolled systemic diseases (e.g., unstable or decompensated respiratory, cardiac, hepatic, or renal diseases) as evaluated by the investigator.
   4. Any unstable systemic disease (including active infection, Grade III hypertension, unstable angina, congestive heart failure, hepatic or renal disease, or metabolic disease).
   5. Inability to take oral medications, requirement for parenteral nutrition, previous surgery affecting absorption, or active gastrointestinal ulceration.
   6. Any significant ocular abnormalities, particularly severe dry eye syndrome, severe dry keratoconjunctivitis, severe exposure keratitis, or other conditions that may increase epithelial damage.
   7. History of known neurologic or psychiatric disorders, including epilepsy or dementia.
5. Insufficient bone marrow reserve or organ function, as indicated by the following laboratory values:

   1. Absolute neutrophil count (ANC) < 1.5 × 10^9/L.
   2. Platelet count < 100 × 10^9/L.
   3. Hemoglobin < 90 g/L (< 9 g/dL).
   4. Alanine aminotransferase (ALT) > 2.5 times the upper limit of normal (ULN).
   5. Aspartate aminotransferase (AST) > 2.5 times ULN.
   6. Total bilirubin > 1.5 times ULN.
   7. Serum creatinine > 1.5 times ULN and creatinine clearance < 60 mL/min (calculated using the Cockcroft-Gault formula); confirmation of creatinine clearance is only required if creatinine is > 1.5 times ULN.
6. Women who are either pregnant or breast-feeding.
7. History of hypersensitivity reactions to any active or inactive components of Aumolertinib or drugs with chemical structures similar to Aumolertinib or in the same class.
8. Patients who may have poor compliance with the study procedures and requirements in the investigator's judgment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-08-15 (Actual); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-10 (Estimated)

PRIMARY OUTCOMES:
ORR (Objective Response Rate) | 3 months.
  ORR (Objective Response Rate) is defined as the proportion of participants who confirmed at least one CR (Complete Response) or PR (Partial response) before disease progression based on Response Evaluation Criteria in Solid Tumors (RECIST)1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
pCR (Pathological Complete Response) | 3 months.
  pCR (Pathological Complete Response) is defined as the proportion of patients in whom no tumor cells are found in all pathological samples after surgical resection following neoadjuvant treatment.
MPR (Major Pathological Response) | 3 months.
  MPR (Major Pathological Response) is defined as the presence of residual tumor of less than 10% on pathological assessment after neoadjuvant treatment-induced tumor regression.
PFS (Progression-Free Survival) | 1 year.
  PFS (Progression-Free Survival) is defined as the time from the first dose of study intervention until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient withdraws from therapy or receives another anti-cancer therapy prior to progression.
OS (Overall Survival) | 1 year.
  OS (Overall Survival) is defined as the time from the initial administration of treatment to the date of death due to any cause. Patients who have not died at the time of statistical analysis will have their survival time censored at the last known date of their survival.

OTHER OUTCOMES:
Changes in EGFR mutation prediction value. | 3 months.
  This analysis observes the changes in the EGFR mutation prediction value of the target lesion diagnosed by AI before and after receiving neoadjuvant treatment with Aumolertinib.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxing He, M.D, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China